CLINICAL TRIAL: NCT05852145
Title: Effect of the Consumption of Beverages Added With Stevia Rebaudiana on Oral pH and Dental Biofilm in Adolescents
Brief Title: Oral Changes With Caloric and no Caloric Sweeteners
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Principal Investigator, Guadalupe Barajas, Principal Investigator, Hospital Infantil de Mexico Federico Gomez
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HIM 2022-049 FF
Record Dates: First submitted 2023-04-09; First posted 2023-05-10 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: pH; Microbiome; Dental Plaque
Keywords: artificial sweetener; stevioside; pH; caries; sucrose; dental biofilm
MeSH Terms: conditions — Dental Plaque | interventions — stevioside; Sucrose; Natural Childbirth

STUDY DESIGN:
Intervention Model Description: A Randomized Crossover Clinical Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: colors will be assigned for each sweetener
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Natural water (Placebo Comparator): 250 ml of natural water should be drunk
  * Salivary pH will be analyzed at 0,5,10,15,30,45 and 60 minutes later
  * Dental biofilm pH will be analyzed at 0,5,10,15,30,45 and 60 minutes later
  * Streptococcus mutans and Streptoccus sobrinus proliferation in dental biofilm ( PCR copies) will be analyzed at 0 and 120 minutes later
  * The relative abundance of Streptococcus mutans and Streptococcus sobrinus in dental biofilm will be analyzed using Amplicon Sequence Variant at 0 and 120 minutes later
  Interventions: Drug: Stevioside; Drug: Sucrose; Other: Natural water
- Stevioside (Experimental): 250 ml of natural water added with 0.1 grams of stevioside should be drunk
  * Salivary pH will be analyzed at 0,5,10,15,30,45 and 60 minutes later
  * Dental biofilm pH will be analyzed at 0,5,10,15,30,45 and 60 minutes later
  * Streptococcus mutans and Streptoccus sobrinus proliferation in dental biofilm ( PCR copies) will be analyzed at 0 and 120 minutes later
  * The relative abundance of Streptococcus mutans and Streptococcus sobrinus in dental biofilm will be analyzed using Amplicon Sequence Variant at 0 and 120 minutes later
  Interventions: Drug: Stevioside; Drug: Sucrose; Other: Natural water
- Sucrose (Active Comparator): 250 ml of natural water added with 25 of sucrose grams with should be drunk.
  * Salivary pH will be analyzed at 0,5,10,15,30,45 and 60 minutes later
  * Dental biofilm pH will be analyzed at 0,5,10,15,30,45 and 60 minutes later
  * Streptococcus mutans and Streptoccus sobrinus proliferation in dental biofilm ( PCR copies) will be analyzed at 0 and 120 minutes later
  * The relative abundance of Streptococcus mutans and Streptococcus sobrinus in dental biofilm will be analyzed using Amplicon Sequence Variant at 0 and 120 minutes later
  Interventions: Drug: Stevioside; Drug: Sucrose; Other: Natural water

INTERVENTIONS:
Drug: Stevioside — 250 ml of natural water added with 0.1 gr. of stevioside should be drunk
  * Salivary pH will be analyzed at 0,5,10,15,30,45 and 60 minutes later
  * Dental biofilm pH will be analyzed at 0,5,10,15,30,45 and 60 minutes later
  * Streptococcus mutans and Strepcotoccus sobrinus proliferation in dental biofilm ( PCR copies) will be analyzed at 0 and 120 minutes later
  * The relative abundance of Streptococcus mutans and Streptococcus sobrinus in dental biofilm will be analyzed using Amplicon Sequence Variant at 0 and 120 minutes later
  Other Names: Non caloric sweetener
Drug: Sucrose — 250 ml of natural water added with 25 gr of sucrose should be drunk
  * Salivary pH will be analyzed at 0,5,10,15,30,45 and 60 minutes later
  * Dental biofilm pH will be analyzed at 0,5,10,15,30,45 and 60 minutes later
  * Streptococcus mutans and Strepcotoccus sobrinus proliferation in dental biofilm ( PCR copies) will be analyzed at 0 and 120 minutes later
  * The relative abundance of Streptococcus mutans and Streptococcus sobrinus in dental biofilm will be analyzed using Amplicon Sequence Variant at 0 and 120 minutes later
  Other Names: Caloric sweetener
Other: Natural water — 250 ml of natural water should be drunk
  * Salivary pH will be analyzed at 0,5,10,15,30,45 and 60 minutes later
  * Dental biofilm pH will be analyzed at 0,5,10,15,30,45 and 60 minutes later
  * Streptococcus mutans and Strepcotoccus sobrinus proliferation in dental biofilm ( PCR copies) will be analyzed at 0 and 120 minutes later
  * The relative abundance of Streptococcus mutans and Streptococcus sobrinus in dental biofilm will be analyzed using Amplicon Sequence Variant at 0 and 120 minutes later

SUMMARY:
The objective of this clinical trial is to compare the effect that the intake of beverages without sweeteners, added with non-caloric sweeteners (stevioside) and caloric sweeteners (sucrose) on oral pH and dental biofilm microbiome in Mexican adolescents.

Participants will drink on different occasions a beverage without sweetener, a beverage added with stevioside or a beverage added with sucrose. The researchers will compare the changes that each one causes in salivary pH, dental biofilm pH, dental biofilm bacterial proliferation and dental biofilm microbiome.

DETAILED DESCRIPTION:
A randomized crossover clinical trial will be conducted including 43 healthy adolescents participants (sample size with alpha=0.05 and beta=0.8 ). The intervention will consist of ingesting 250 mL of natural water (pH 7.1) in the first meeting, in subsequent meetings the natural water will be added with 1) 0.1 gr. of stevioside or 2) 25 gr. of sucrose. The washout period between interventions will be 1 week.

Participants will be informed of potential risks and those who sign the informed consent and complete the inclusion criteria will be randomized in a triple-blind manner.

The data will be collected in a special format including previous conditions, identification (age and sex) and possible adverse effects. If any possible adverse effect occurs, it will be notified to the research team to determine the changes.

* To determine the pH, saliva and dental biofilm samples will be obtained and analyzed using a HANNA potentiometer.
* To determine the bacterial proliferation, samples of dental biofilm will be obtained and the number of copies of Streptococcus mutans (S. mutans) and Streptococcus sobrinus (S. sobrinus) will be analyzed by polymerase reaction technique (PCR) of the 16S ribosomal gene fragment.
* To analyze dental biofilm microbiome, 11 of the 43 participants will be randomized for. Genetic sequencing will be performed and the amplicon Sequence Variants (ASVs) of S. mutans and S. sobrinus will be compared.

The data will be collected at a time indicated by a stopwatch and carried out by two verifiers.

The statistical analysis will be done according to the type of variable, these will be described with mean and standard deviation or frequencies and percentages. The pH will be compared by ANOVA analysis and adjusted by Bonferroni correction. Bacterial proliferation will be analyzed by Kruskal Wallis test. Statistical Package for the Social Sciences (SPSS) v. 22 program will be used considering p value ≤ 0.05. For the microbiome, the Amplicon Sequence Variants (ASVs) will be analyzed. Non-parametric multivariate analysis of variance and an analysis of similarities will be used. The p values will be calculated, identifying those that have differences in bacterial communities between the groups using the Genius (V3) software.

ELIGIBILITY:
Inclusion Criteria:

* Habitual consumption of soft drinks
* Decayed, Missing, and Filled Teeth (DMF) index of at least 3 (considering as caries those lesions that are visible without the tooth needing to be dry)
* Agree to participate in the study and sign informed consent
* Parents sign informed consent
* Any nutritional condition

Exclusion Criteria:

* Orthodontic treatment
* Topical application of fluoride during the last 3 months
* Having a motor disability that interfered with tooth brushing
* Xerostomia
* Antibiotic therapy during the study period
* Periodontal infections

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Mean salivary pH with natural water | 0 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water | 5 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water | 10 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water | 15 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water | 30 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water | 45 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water | 60 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water added with 25 gr of sucrose | 0 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water added with 25 gr of sucrose | 5 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water added with 25 gr of sucrose | 10 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water added with 25 gr of sucrose | 15 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water added with 25 gr of sucrose | 30 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water added with 25 gr of sucrose | 45 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water added with 25 gr of sucrose | 60 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water added with 0.1 gr of stevioside | 0 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water added with 0.1 gr of stevioside | 5 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water added with 0.1 gr of stevioside | 10 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water added with 0.1 gr of stevioside | 15 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water added with 0.1 gr of stevioside | 30 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water added with 0.1 gr of stevioside | 45 minutes
  Logarithm of hydrogen ion concentration
Mean salivary pH with natural water added with 0.1 gr of stevioside | 60 minutes
  Logarithm of hydrogen ion concentration

SECONDARY OUTCOMES:
Mean dental biofilm pH with natural water | 0 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water | 5 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water | 10 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water | 15 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water | 30 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water | 45 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water | 60 minutes
  Logarithm of hydrogen ion concentration
Mean Mean dental biofilm pH with natural water added with 25 gr of sucrose | 0 minutes
  Logarithm of hydrogen ion concentration
Mean Mean dental biofilm pH with natural water added with 25 gr of sucrose | 5 minutes
  Logarithm of hydrogen ion concentration
Mean Mean dental biofilm pH with natural water added with 25 gr of sucrose | 10 minutes
  Logarithm of hydrogen ion concentration
Mean Mean dental biofilm pH with natural water added with 25 gr of sucrose | 15 minutes
  Logarithm of hydrogen ion concentration
Mean Mean dental biofilm pH with natural water added with 25 gr of sucrose | 30 minutes
  Logarithm of hydrogen ion concentration
Mean Mean dental biofilm pH with natural water added with 25 gr of sucrose | 45 minutes
  Logarithm of hydrogen ion concentration
Mean Mean dental biofilm pH with natural water added with 25 gr of sucrose | 60 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water added with 0.1 gr stevioside | 0 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water added with 0.1 gr stevioside | 5 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water added with 0.1 gr stevioside | 10 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water added with 0.1 gr stevioside | 15 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water added with 0.1 gr stevioside | 30 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water added with 0.1 gr stevioside | 45 minutes
  Logarithm of hydrogen ion concentration
Mean dental biofilm pH with natural water added with 0.1 gr stevioside | 60 minutes
  Logarithm of hydrogen ion concentration

OTHER OUTCOMES:
Dental biofilm proliferation with natural water | 0 minutes
  S. mutans and S. sobrinus number of copies
Dental biofilm proliferation with natural water | 120 minutes
  S. mutans and S. sobrinus number of copies
Dental biofilm proliferation with natural water added with 25 gr of sucrose | 0 minutes
  S. mutans and S. sobrinus number of copies
Dental biofilm proliferation with natural water added with 25 gr of sucrose | 120 minutes
  S. mutans and S. sobrinus number of copies
Dental biofilm proliferation with natural water added with 0.1 gr of stevioside | 0 minutes
  S. mutans and S. sobrinus number of copies
Dental biofilm proliferation with natural water added with 0.1 gr stevioside | 120 minutes
  S. mutans and S. sobrinus number of copies
Microbiome abundance with natural water | 0 minutes
  S. mutans and S. sobrinus amplicon sequence variant
Microbiome abundance with natural water | 120 minutes
  S. mutans and S. sobrinus amplicon sequence variant
Microbiome abundance with natural water added with 25 gr sucrose | 0 minutes
  S. mutans and S sobrinus Amplicon sequence variant
Microbiome abundance with natural water added 25 gr of sucrose | 120 minutes
  S. mutans and S. sobrinus amplicon sequence variant
Microbiome abundance with natural water added with 0.1 gr. of stevioside. | 0 minutes
  S. mutans and S. sobrinus amplicon sequence variant
Microbiome abundance with natural water added with 0.1 gr. of stevioside. | 120 minutes
  S. mutans and S sobrinus amplicon sequence variant

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Barajas, MsC, Principal Investigator — Children´s Hospital Federico Gómez. México
Locations (1):
- Hospital Infantil de México Federico Gomez, Mexico City, Cuahutemoc, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Yes: There is a plan to make Individual Participant Data (IPD) Sharing Statement.
Supporting Information: SAP, ICF
Time Frame: At the time of manuscript publication
Access Criteria: Asking for email
URL: https://docs.google.com/spreadsheets/d/1LbhMW8PgO2wFkcQ-2V59iOXrU357_i9lVocikpc6J8s/edit?usp=sharing

REFERENCES:
- [Background] Struzycka I. The oral microbiome in dental caries. Pol J Microbiol. 2014;63(2):127-35. PMID 25115106
- [Background] Edelstein BL. The dental caries pandemic and disparities problem. BMC Oral Health. 2006 Jun 15;6 Suppl 1(Suppl 1):S2. doi: 10.1186/1472-6831-6-S1-S2. PMID 16934119
- [Background] Moradi G, Mohamadi Bolbanabad A, Moinafshar A, Adabi H, Sharafi M, Zareie B. Evaluation of Oral Health Status Based on the Decayed, Missing and Filled Teeth (DMFT) Index. Iran J Public Health. 2019 Nov;48(11):2050-2057. PMID 31970104
- [Background] Carvalho RN, Letieri ADS, Vieira TI, Santos TMPD, Lopes RT, Neves AA, Pomarico L. Accuracy of visual and image-based ICDAS criteria compared with a micro-CT gold standard for caries detection on occlusal surfaces. Braz Oral Res. 2018 Jul 10;32:e60. doi: 10.1590/1807-3107bor-2018.vol32.0060. PMID 29995065
- [Background] Skrivele S, Care R, Berzina S, Kneist S, de Moura-Sieber V, de Moura R, Borutta A, Maslak E, Tserekhava T, Shakovets N, Wagner M. Caries and its risk factors in young children in five different countries. Stomatologija. 2013;15(2):39-46. PMID 24037301
- [Background] Aamodt K, Reyna-Blanco O, Sosa R, Hsieh R, De la Garza Ramos M, Garcia Martinez M, Orellana MF. Prevalence of caries and malocclusion in an indigenous population in Chiapas, Mexico. Int Dent J. 2015 Oct;65(5):249-55. doi: 10.1111/idj.12177. Epub 2015 Sep 18. PMID 26382724
- [Background] Irigoyen ME, Mejia-Gonzalez A, Zepeda-Zepeda MA, Betancourt-Linares A, Lezana-Fernandez MA, Alvarez-Lucas CH. Dental caries in Mexican schoolchildren: a comparison of 1988-1989 and 1998-2001 surveys. Med Oral Patol Oral Cir Bucal. 2012 Sep 1;17(5):e825-32. doi: 10.4317/medoral.18008. PMID 22549683
- [Background] Garcia-Cortes JO, Mejia-Cruz JA, Medina-Cerda E, Orozco-De la Torre G, Medina-Solis CC, Marquez-Rodriguez S, Navarrete-Hernandez Jde J, Islas-Granillo H. [Experience, prevalence, severity, treatment needs for dental caries and care index in Mexican adolescents and young adults]. Rev Invest Clin. 2014 Nov-Dec;66(6):505-11. Spanish. PMID 25729867
- [Background] Krzysciak W, Pluskwa KK, Piatkowski J, Krzysciak P, Jurczak A, Koscielniak D, Skalniak A. The usefulness of biotyping in the determination of selected pathogenicity determinants in Streptococcus mutans. BMC Microbiol. 2014 Aug 5;14:194. doi: 10.1186/1471-2180-14-194. PMID 25096795
- [Background] Mathur MR, Tsakos G, Millett C, Arora M, Watt R. Socioeconomic inequalities in dental caries and their determinants in adolescents in New Delhi, India. BMJ Open. 2014 Dec 12;4(12):e006391. doi: 10.1136/bmjopen-2014-006391. PMID 25500618
- [Background] Humphrey SP, Williamson RT. A review of saliva: normal composition, flow, and function. J Prosthet Dent. 2001 Feb;85(2):162-9. doi: 10.1067/mpr.2001.113778. PMID 11208206
- [Background] Kaur A, Kwatra KS, Kamboj P. Evaluation of non-microbial salivary caries activity parameters and salivary biochemical indicators in predicting dental caries. J Indian Soc Pedod Prev Dent. 2012 Jul-Sep;30(3):212-7. doi: 10.4103/0970-4388.105013. PMID 23263424
- [Background] He J, Li Y, Cao Y, Xue J, Zhou X. The oral microbiome diversity and its relation to human diseases. Folia Microbiol (Praha). 2015 Jan;60(1):69-80. doi: 10.1007/s12223-014-0342-2. Epub 2014 Aug 23. PMID 25147055
- [Background] Koo H, Falsetta ML, Klein MI. The exopolysaccharide matrix: a virulence determinant of cariogenic biofilm. J Dent Res. 2013 Dec;92(12):1065-73. doi: 10.1177/0022034513504218. Epub 2013 Sep 17. PMID 24045647
- [Background] Foglio-Bonda PL, Brilli K, Pattarino F, Foglio-Bonda A. Salivary flow rate and pH in patients with oral pathologies. Eur Rev Med Pharmacol Sci. 2017 Jan;21(2):369-374. PMID 28165549
- [Background] Ilie O, van Turnhout AG, van Loosdrecht MC, Picioreanu C. Numerical modelling of tooth enamel subsurface lesion formation induced by dental plaque. Caries Res. 2014;48(1):73-89. doi: 10.1159/000354123. Epub 2013 Nov 14. PMID 24248036
- [Background] Pandey P, Reddy NV, Rao VA, Saxena A, Chaudhary CP. Estimation of salivary flow rate, pH, buffer capacity, calcium, total protein content and total antioxidant capacity in relation to dental caries severity, age and gender. Contemp Clin Dent. 2015 Mar;6(Suppl 1):S65-71. doi: 10.4103/0976-237X.152943. PMID 25821379
- [Background] Escobar E, Piedrahita M, Gregory RL. Growth and viability of Streptococcus mutans in sucrose with different concentrations of Stevia rebaudiana Bertoni. Clin Oral Investig. 2020 Sep;24(9):3237-3242. doi: 10.1007/s00784-020-03197-5. Epub 2020 Mar 18. PMID 32189073
- [Background] Brambilla E, Cagetti MG, Ionescu A, Campus G, Lingstrom P. An in vitro and in vivo comparison of the effect of Stevia rebaudiana extracts on different caries-related variables: a randomized controlled trial pilot study. Caries Res. 2014;48(1):19-23. doi: 10.1159/000351650. Epub 2013 Nov 6. PMID 24216624
- [Background] Behjati S, Tarpey PS. What is next generation sequencing? Arch Dis Child Educ Pract Ed. 2013 Dec;98(6):236-8. doi: 10.1136/archdischild-2013-304340. Epub 2013 Aug 28. PMID 23986538